CLINICAL TRIAL: NCT01006720
Title: Dose Finding Study for Sugammadex and Neostigmine at Residual Neuromuscular Blockade (T4/T1 = 0.2)
Brief Title: Sugammadex and Neostigmine at Residual Neuromuscular Blockade
Acronym: SUNDRO20
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: SUNDRO20; EudraCT number 2009-013499-29
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Residual Neuromuscular Block (TOF-ratio of 0.2)
Keywords: Residual neuromuscular block; post-operative residual curarization; PORC; sugammadex; neostigmine
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex; Neostigmine; Sodium Chloride

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (11):
- Sgx 0.25: Sugammadex group: Different doses of sugammadex for reversal of shallow neuromuscular blockade
  Interventions: Drug: Sugammadex
- Sgx 0.5: Sugammadex group: Different doses of sugammadex for reversal of shallow neuromuscular blockade
  Interventions: Drug: Sugammadex
- Sgx 0.75: Sugammadex group: Different doses of sugammadex for reversal of shallow neuromuscular blockade
  Interventions: Drug: Sugammadex
- Sgx 1.0: Sugammadex group: Different doses of sugammadex for reversal of shallow neuromuscular blockade
  Interventions: Drug: Sugammadex
- Sgx 1.25: Sugammadex group: Different doses of sugammadex for reversal of shallow neuromuscular blockade
  Interventions: Drug: Sugammadex
- Neo 10: Neostigmine group: Different doses of neostigmine for reversal of shallow neuromuscular blockade
  Interventions: Drug: Neostigmine
- Neo 25: Neostigmine group: Different doses of neostigmine for reversal of shallow neuromuscular blockade
  Interventions: Drug: Neostigmine
- Neo 40: Neostigmine group: Different doses of neostigmine for reversal of shallow neuromuscular blockade
  Interventions: Drug: Neostigmine
- Neo 55: Neostigmine group: Different doses of neostigmine for reversal of shallow neuromuscular blockade
  Interventions: Drug: Neostigmine
- Neo 70: Neostigmine group: Different doses of neostigmine for reversal of shallow neuromuscular blockade
  Interventions: Drug: Neostigmine
- Saline: Saline group: Saline as placebo
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Sugammadex — Single intravenous injection of either:
  Sugammadex 0.25 mg/kg (Sgx 0.25) Sugammadex 0.5 mg/kg (Sgx 0.5) Sugammadex 0.75 mg/kg (Sgx 0.75) Sugammadex 1.0 mg/kg (Sgx 1.0) Sugammadex 1.25 mg/kg (Sgx 1.25)
  Groups: Sgx 0.25; Sgx 0.5; Sgx 0.75; Sgx 1.0; Sgx 1.25
Drug: Neostigmine — Neostigmine 10 µg/kg (Neo 10) Neostigmine 25 µg/kg (Neo 25) Neostigmine 40 µg/kg (Neo 40) Neostigmine 55 µg/kg (Neo 55) Neostigmine 70 µg/kg (Neo 70)
  Groups: Neo 10; Neo 25; Neo 40; Neo 55; Neo 70
Drug: Saline — Saline 0.9% (Saline)
  Groups: Saline

SUMMARY:
This study is designed to compare recovery times after reversal of a residual neuromuscular block (TOF-ratio 0.2) with different doses of either neostigmine or sugammadex.

DETAILED DESCRIPTION:
Muscle relaxants are integral part of modern anesthesia. They optimize intubating conditions, reduce laryngeal trauma and improve operating conditions. Drawback is a possible pharmacological (muscle relaxing) effect of these drugs beyond the end of the operation (i.e. post-operative residual curarization: PORC). Reportedly about 30% of all patients who received muscle relaxants show signs of PORC when arriving in the post-anesthesia care unit. PORC comprises the risk of impaired post-operative fine motor and coordinative skills with a possible impairment of swallowing pharyngeal secretions with an increased risk of aspiration after extubation. Possible deleterious effects of this could be pneumonia, bronchitis, myocardial infarction, cardiac insufficiency, stroke or re-operation.

In order to avoid PORC patients with residual neuromuscular block receive a muscle relaxant antagonist from the anesthesiologist at the end of the operation. However, these drugs (neostigmine, pyridostigmine, etc.) from the class of cholinesterase inhibitors have unwanted effects such as bradycardia, increased gastro-intestinal motility, post-operative nausea and vomiting, salivation etc. To decrease these unwanted side effects cholinesterase inhibitors have to be given in combination with parasympatholyics e.g. atropine or glycopyrrolate with their own spectrum of unwanted side effects.

From October 2008 on, Sugammadex, a completely new reversal drug was introduced in to clinical practice. Sugammadex, is a modified γ-cyclodextrine able to specifically bind rocuronium (a steroidal muscle relaxant). The complex is eliminated via the kidneys. However, all studies so far have focussed on reversal of profound or deep neuromuscular blockade. This study is designed to compare recovery times after reversal of a residual neuromuscular block (TOF-ratio 0.2) with different doses of either the neostigmine or sugammadex.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA physical status I - III
* Patients over 18 years
* Patients scheduled for general anesthesia with intubation using rocuronium
* Patients having given informed consent to the study

Exclusion Criteria:

* Anatomic and functional malformations with expected difficult intubation
* Known or suspected neuromuscular disease
* Significant hepatic or renal dysfunction
* Known or suspected history or family history of disposition to malignant hyperthermia
* Known or suspected allergy towards sugammadex, anesthetics, muscle relaxants, or other drugs used for general anesthesia
* Use of drugs that interfere with muscle relaxants
* Patients, included in another trial within the last 30 days
* Patients, with legal guidant
* Patients with contraindication towards the use of Sugammadex, neostigmine or glycopyrrolate
* Patients, which have already participated in a sugammadex trial
* Pregnant women (exclusion of pregnancy: postmenopausal status, negative β- HCG screen, status post tubal ligation)
* Breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving rocuronium for neuromuscular blockade under general anesthesia
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time to TOF-ratio 0.9 following the investigational drug | Regular anesthesia time, approximately 1.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Heidrun Fink, PD Dr., MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Ismaninger Str. 22, 81675 München
Locations (1):
- Klinik für Anaesthesiologie, Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- [Background] Puhringer FK, Rex C, Sielenkamper AW, Claudius C, Larsen PB, Prins ME, Eikermann M, Khuenl-Brady KS. Reversal of profound, high-dose rocuronium-induced neuromuscular blockade by sugammadex at two different time points: an international, multicenter, randomized, dose-finding, safety assessor-blinded, phase II trial. Anesthesiology. 2008 Aug;109(2):188-97. doi: 10.1097/ALN.0b013e31817f5bc7. PMID 18648227
- [Background] Flockton EA, Mastronardi P, Hunter JM, Gomar C, Mirakhur RK, Aguilera L, Giunta FG, Meistelman C, Prins ME. Reversal of rocuronium-induced neuromuscular block with sugammadex is faster than reversal of cisatracurium-induced block with neostigmine. Br J Anaesth. 2008 May;100(5):622-30. doi: 10.1093/bja/aen037. Epub 2008 Apr 2. PMID 18385265
- [Derived] Kaufhold N, Schaller SJ, Stauble CG, Baumuller E, Ulm K, Blobner M, Fink H. Sugammadex and neostigmine dose-finding study for reversal of residual neuromuscular block at a train-of-four ratio of 0.2 (SUNDRO20)dagger, Br J Anaesth. 2016 Feb;116(2):233-40. doi: 10.1093/bja/aev437. PMID 26787792